CLINICAL TRIAL: NCT03566225
Title: Combined Pioglitazone and Clomophene Citrate Versus Combined Metformin and Clomiphene Citrate as First Treatment in Infertile Women With Polycystic Ovary Syndrome
Brief Title: Pioglitazone Versus Metformin as First Treatment in Infertile Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelbadea Ali Salih, Cairo, Ain Shams University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AinShamaU
Record Dates: First submitted 2018-05-26; First posted 2018-06-25 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Pioglitazone
MeSH Terms: interventions — Pioglitazone; Metformin; Clomiphene

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Pioglitazone in adose 30 mg tablet will be administered dialy+ clomiphene citrate as ovulation induction
  Interventions: Drug: Pioglitazone; Drug: Clomiphene Citrate
- Group B (Placebo Comparator): Metformin in adose 1500 mg dialy will be administered + clomiphene citrate
  Interventions: Drug: Metformin; Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Pioglitazone — Insulin sensitizing agents
  Other Names: Glustazon
  Arms: Group A
Drug: Metformin — Insulin sensitizing agent
  Other Names: Cidophage
  Arms: Group B
Drug: Clomiphene Citrate — Induction drug
  Other Names: Clomid

SUMMARY:
Participants with PCOS will be divided into two groups then each group will randomly recieve one of the following treatment

1. metformin will be adminstered in adose of 500 mg 3 times daily for 3 months to group B.
2. pioglitazone will be administered in adose of 30 mg dialy for 3 months to group A.
3. Induction of ovulation by clomiphene citate 50 mg tablets to all participants

DETAILED DESCRIPTION:
Participants with PCOS will be divided into two groups then each group will randomly recieve one of the following treatment

1. metformin will be adminstered in adose of 500 mg 3 times daily for 3 months to group B.
2. pioglitazone will be administered in adose of 30 mg dialy for 3 months to group A.
3. Induction of ovulation by clomiphene citate 50 mg tablets once or twice dialy 12hours apart starting from the 3rd day of menstrual cycle and continue for five days during treatment with insulin sensitizing agents to group A and B.

Participants with oligomenorrhea will recieve two tablets of noreththisterone 5 mg tab every 12 hours for 5 days to allow for withdrawal bleeding before start ovulation induction

ELIGIBILITY:
Inclusion Criteria:

* women age 20_35
* BMI 18_29.9
* Women with PCOS(diagnosed by using Rotterdam criteria
* Infertility is cause for seeking tfeatment

Exclusion Criteria:

* Causes of infertility other than PCOS.
* patient refusal.
* Contraindication of any of the drugs used in the study
* Cause of oligo/anovulation other than PCOS
* Current or previous (within the last six month) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetics, antiobesity drugs or other hormonal drugs.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 3 months
  Pregnancy rate diagnosed by U/S at five weeks after missed menses

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Salih, Resident, Principal Investigator — AinShams University
Locations (1):
- Ain Shams Univerisity, Cairo, Egypt